CLINICAL TRIAL: NCT04027452
Title: Electroconvulsive Therapy for Traumatic Memories: A Randomized Controlled Clinical Trial
Brief Title: Electroconvulsive Therapy for Traumatic Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Albert Wong, Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 063/2015
Record Dates: First submitted 2019-07-04; First posted 2019-07-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Post Traumatic Stress Disorder; Depression
Keywords: electroconvulsive therapy; post traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Traumatic memory reactivation (Experimental): Audio recording of traumatic memory that triggers symptoms of PTSD, anxiety, depression, played before each ECT treatment.
  Interventions: Behavioral: Traumatic memory reactivation
- Neutral memory reactivation (Placebo Comparator): Audio recording of neutral (non-traumatic) memory played before each ECT treatment.
  Interventions: Behavioral: Neutral memory reactivation

INTERVENTIONS:
Behavioral: Traumatic memory reactivation — 125 word long "exposure scripts" of their traumatic memory recorded in a neutral tone. All recordings will be approximately 30 seconds in length and the traumatic script will include five of the physical symptoms related to the memory as described by the patient. The script recording is preceded with short instructions for the subject to concentrate on the script and to imagine the described experience for additional 30 seconds right after the script until a short beep sounds. When the participant enters the treatment room, they will be handed an MP3 player with the audio recording. The patient will have several minutes to listen to the recording while the standard pre-ECT procedures are conducted. The participant will listen to the recording prior to each of their ECT treatments for the duration of their acute treatment course.
  Arms: Traumatic memory reactivation
Behavioral: Neutral memory reactivation — 125 word long "exposure scripts" of a neutral (non-traumatic) memory recorded in a neutral tone. All recordings will be approximately 30 seconds in length and the traumatic script will include five of the physical symptoms related to the memory as described by the patient. The script recording is preceded with short instructions for the subject to concentrate on the script and to imagine the described experience for additional 30 seconds right after the script until a short beep sounds. When the participant enters the treatment room, they will be handed an MP3 player with the audio recording. The patient will have several minutes to listen to the recording while the standard pre-ECT procedures are conducted. The participant will listen to the recording prior to each of their ECT treatments for the duration of their acute treatment course.
  Arms: Neutral memory reactivation

SUMMARY:
This study will investigate whether ECT treatment can reduce the effect of traumatic memories if those memories are recalled immediately prior to the ECT sessions. Participants will be randomized to either a recall of a traumatic memory or a neutral non-traumatic memory prior to their ECT sessions.

DETAILED DESCRIPTION:
Traumatic events contribute to the genesis of disorders such as post-traumatic stress disorder (PTSD) and depression, and memories of the event can cause ongoing distress. Short-term episodic memories are encoded by the hippocampus and gradually become consolidated through reciprocal connections with the cortex, resulting in long-term memories being stored in a distributed network throughout the cerebral cortex. There are no effective treatments currently for specifically targeting traumatic memories and reducing the distress they cause.

ECT is the most effective treatment for improving mood in patients with depression and there is new evidence emerging that suggests ECT can also improve PTSD symptoms independently of co-morbid depression. In addition, the main side-effect of ECT is memory loss, specifically for autobiographical details surrounding the course of ECT, but not typically affecting long-term episodic memory, nor procedural memories. Memories stored in the hippocampus are vulnerable to disruption by ECT because they rely on synaptic changes that are mediated by relatively unstable modifications in AMPA receptor and metabotropic glutamate receptor density. The investigators propose to exploit this feature of ECT, which normally is considered an undesirable side-effect of treatment, in an attempt to selectively reduce traumatic memories and the distress associated with them.

The investigators propose to recruit patients referred for ECT for treatment-resistant depression, who also have traumatic memories that are causing distress. These patients will be asked to write two narratives, one of the traumatic memory, and the other of a trivial, non-traumatic remote event. Patients will then be asked to listen to an audio recording of either the traumatic memory or the neutral memory (control group) immediately before their ECT sessions. The severity of the traumatic memory related symptoms will be assessed before and after the course of ECT using the Modified PTSD Symptom Scale (MPSS-SR) and the Clinician Administered PTSD Scale for DSM-5 (CAPS-5). Data will be analyzed by comparing the change in overall MPSS-SR scores and CAPS-5 scores pre- and post-ECT between the experimental and control groups. Physiological data will also be collected at each ECT session during the time the participant is listening to the audio recordings. Heart rate and skin conductance will be measured prior to and during listening of the traumatic or non-traumatic memory, in order to determine if there is a change associated with a stress response, and whether this response normalizes in association with reduction of PTSD symptoms with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred and accepted for ECT treatment at CAMH
2. Presence of traumatic memories
3. Able to write about their traumatic experience(s)
4. Capable of informed consent to participate in this study
5. Age 18 or greater
6. MPSS-SR re-experiencing score (items 1-4, 17) ≥ 20

Exclusion Criteria:

1. History of neurological or developmental disorder, including seizures
2. ECT treatment already started

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Modified PTSD Symptom Scale (MPSS-SR) score | Baseline, after ECT treatment course (an average of 4 weeks), and at 3 month follow up
  17-item self-report measure that assesses the DSM-III-R symptoms of PTSD. Score range from 0-119, higher score indicates greater PTSD symptom severity.
Change in Clinician Administered PTSD Scale for DSM-5 (CAPS-5) score | Baseline, after ECT treatment course (an average of 4 weeks), and at 3 month follow up
  30-item semi structured interview that is used to index of PTSD severity and assess PTSD symptoms over the past week. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, and impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, and features for the dissociative subtype (depersonalization and derealization). Administration requires identification of an index traumatic event to serve as the basis for symptom inquiry. Symptom severity scores range from 0 to 80, higher score indicates greater PTSD symptom severity.

SECONDARY OUTCOMES:
Change in heart rate | Change of heart rate from 0-30 seconds of the audio recording to heart rate from 90-120 seconds of the audio recording.
  Heart rate change before and after listening to script of traumatic or neutral memory
Skin conductance | Change of skin conductance from 0-30 seconds of the audio recording to skin conductance from 90-120 seconds of the audio recording.
  Skin conductance change before and after listening to script of traumatic or neutral memory
Change in The Quick Inventory of Depressive Symptomatology (Self-Report) | Baseline, after ECT treatment course (an average of 4 weeks), and at 3 month follow up
  Self report scale of depressive symptoms. Scores range from 0-27, higher score indicates greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Albert HC Wong, MD, FRCPC, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang VM, Trought K, Gicas KM, Kozak M, Josselyn SA, Daskalakis ZJ, Blumberger DM, Voineskos D, Knyahnytska Y, Pasricha S, Chung Y, Zhou Y, Isserles M, Wong AHC. Electroconvulsive therapy with a memory reactivation intervention for post-traumatic stress disorder: A randomized controlled trial. Brain Stimul. 2021 May-Jun;14(3):635-642. doi: 10.1016/j.brs.2021.03.015. Epub 2021 Mar 27. PMID 33785406

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04027452/Prot_SAP_000.pdf